CLINICAL TRIAL: NCT00897975
Title: Red Yeast Rice and Phytosterols Versus Red Yeast Rice and Placebo for the Treatment of Hyperlipidemia in Patients With Statin Intolerance: A Multi-Center Randomized Double-blind Study
Brief Title: Red Yeast Rice and Phytosterols In Statin Intolerance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chestnut Hill Health System (Other)
Responsible Party: David Becker, MD, Chestnut Hill Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWA00005390 Chestnut HillHC
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2009-11

CONDITIONS: Hyperlipidemia
Keywords: statin associated myalgias; hyperlipidemia; red yeast rice; phytosterols; therapeutic lifestyle changes; compliance
MeSH Terms: conditions — Hyperlipidemias; Patient Compliance | interventions — red yeast rice; Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- red yeast rice (RYR) plus phytosterol (Experimental): arm will take red yeast rice and phytosterol supplement
  Interventions: Dietary Supplement: red yeast rice; Drug: phytosterol
- red yeast rice plus placebo (Placebo Comparator)
  Interventions: Dietary Supplement: red yeast rice; Drug: placebo
- TLC plus red yeast rice plus placebo (Active Comparator): subjects attend 12 week therapeutic lifestyle program and take above supplement
  Interventions: Dietary Supplement: red yeast rice; Behavioral: therapeutic lifestyle program; Drug: placebo
- TLC plus RYR plus phytosterol (Experimental): Therapeutic lifestyle program for 12 weeks plus red yeast rice plus phytosterol
  Interventions: Dietary Supplement: red yeast rice; Drug: phytosterol; Behavioral: therapeutic lifestyle program

INTERVENTIONS:
Dietary Supplement: red yeast rice — 600 mg 3 capsules bid
Drug: phytosterol — phytosterol 450 mg 2 tabs bid with food
  Arms: TLC plus RYR plus phytosterol; red yeast rice (RYR) plus phytosterol
Behavioral: therapeutic lifestyle program — TLC - 12 weeks
  Arms: TLC plus RYR plus phytosterol; TLC plus red yeast rice plus placebo
Drug: placebo — placebo
  Arms: TLC plus red yeast rice plus placebo; red yeast rice plus placebo

SUMMARY:
Red yeast rice may be useful to lower cholesterol, especially in a population of patients who cannot tolerate traditional therapy with statins.

The addition of an over-the-counter phytosterol to red yeast rice may offer additional lipid lowering benefits when compared to red yeast rice alone.

These supplements will be given to all participants. Up to one-half will enroll in a lifestyle intervention program called Change of Heart and will be compared to patients who do not participate in the program. The study will last one year.

DETAILED DESCRIPTION:
Although recent studies have shown that red yeast rice is an effective therapy in the treatment of hyperlipidemia, additional supplements may be required to lower cholesterol to levels that have been associated with decreased coronary events. Specifically a target has been to lower low-density lipoprotein-C (LDL-C) to levels below 100 mg/dl. Red yeast rice has been found to be effective in lowering cholesterol in the context of the Change of Heart Program, where participants are encouraged to make significant lifestyle changes. This has been documented in two recent trials that we have published in the past year in the Mayo Clinic Proceedings (July 2008) and The Annals of Internal Medicine (in press). Clinically, we have found it necessary to add a phytosterol supplement to red yeast rice to lower LDL-C levels below 100 mg/dl. There has been a great deal of interest in phytosterols in both the lay and medical press in the past several years. This over the counter supplement lowers cholesterol by acting in the intestine to decrease the absorption of cholesterol. As it is not absorbed, there have not been any reports of significant side effects. The purpose of this study is to examine the lipid lowering effects of red yeast rice with and without adding a phytosterol. Some participants will attend the Change of Heart Program and take these supplements. Another group of participants will take the same supplements, with their usual medical care, but not enroll in the Change of Heart Program. The study will last one year, and participants will have been intolerant of statins in the past.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age > 21
* LDL > 100 and physician suggestion to take statin
* Subject complains of muscle weakness or aching which he/she or his/her physician feels may be attributable to statin therapy
* Having stopped a statin drug for personal reasons and not willing to restart this medication
* Refusal to take a statin as prescribed by personal physician
* CPK < 400
* Not taking any cholesterol lowering medication, red yeast rice extract or a phytosterol product for at least 1 month prior to initiation of trial
* Ability to exercise without physical restrictions
* Ability to attend 12 week consecutive Change of Heart lifestyle education sessions
* Liver function studies normal at baseline
* Subject willing to remain off the dietary supplement CoQ10 for duration of trial
* TSH must be normal

Exclusion Criteria:

* A history of muscle damage (CPK > 400 IU) on statin therapy
* Any active cardiac problem including chest pain, angina, shortness of breath with minimal activity, or unstable angina/acute coronary syndrome within one year
* Known intolerance to one of the study drugs
* Physical limitation preventing aerobic exercise program, such as severe arthritis, peripheral vascular disease, congestive heart failure, or symptom limiting pulmonary disease
* Uncontrolled hypertension (defined as SBP > 180 mmHg or DBP > 100 mmHg
* Heart attack, bypass surgery, or angioplasty/stent within 1 year of study
* Triglyceride level more than 400 mg/dl
* Underlying musculoskeletal disorder preventing muscle testing
* Taking other medicines including: cyclosporine, erythromycin or other macrolide antibiotics; fluconazole; niacin; fibrates; or > 16 oz. of grapefruit juice daily

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol levels | one year

SECONDARY OUTCOMES:
myalgia compared to prior statin usage | one year
other lipoprotein levels | one year
weight loss in TLC program vs. baseline | one year

CONTACTS AND LOCATIONS:
Overall Officials: David J Becker, MD, Principal Investigator — Chestnut Hill Heathcare
Locations (2):
- United States (2):
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Chestnut Hill Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Becker DJ, French B, Morris PB, Silvent E, Gordon RY. Phytosterols, red yeast rice, and lifestyle changes instead of statins: a randomized, double-blinded, placebo-controlled trial. Am Heart J. 2013 Jul;166(1):187-96. doi: 10.1016/j.ahj.2013.03.019. Epub 2013 Apr 30. PMID 23816039